CLINICAL TRIAL: NCT03700567
Title: Safety and Efficacy of Low Temperature Contrast for the Treatment of PCI-related Myocardial Injury in Patients With Unstable Angina Pectoris (LOTA-I)
Brief Title: Safety and Efficacy of Low Temperature Contrast in UAP Patients During PCI (LOTA-I)
Acronym: LOTA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20180713-03
Record Dates: First submitted 2018-09-29; First posted 2018-10-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Unstable Angina Pectoris
Keywords: low temperature; contrast; PCI-related myocardial injury
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low temperature contrast (Experimental): A total of 220 patients are assigned to low temperature contrast group after randomization schedule.
  Interventions: Other: low temperature contrast
- room temperature contrast (No Intervention): A total of 220 patients are assigned to room temperature contrast group after randomization schedule.

INTERVENTIONS:
Other: low temperature contrast — UAP patients undergoing PCI were performed with low temperature contrast. The investigators used thermal insulation equipment to keep contrast at 5℃. The EKG and blood pressure were monitored during the PCI procedure. After PCI, the investigators monitored levels of myocardial injury biomarkers for 3 days every 8 hours.
  Arms: low temperature contrast

SUMMARY:
Percutaneous coronary intervention (PCI) has become one of the main treatments for rapid recovery of revascularization in patients with coronary heart disease (CHD). PCI has some advantages, such as easy operation, small trauma and rapid recovery. It can significantly improve myocardial ischemic symptom and reduce the incidence of cardiovascular adverse events in CHD patients. However, many studies have found that the incidence of PCI-related myocardial injury is relatively high, and affect the efficacy of PCI and prognosis in patients with unstable angina pectoris (UAP). A meta-analysis of a total of 7578 patients with UAP from 15 studies who underwent PCI was found to have a 28.7% increase in myocardial biomarkers after PCI. The objective of this randomized control trial is to gain a clinical insight on the use of low temperature contrast for the treatment of PCI-related myocardial injury in UAP patients. The primary objective is assess efficacy and safety of low temperature contrast for the treatment of PCI-related myocardial injury in UAP patients.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the change in levels of myocardial injury biomarkers (such as TNI and CK-MB) between low temperature contrast group and room temperature contrast group. Based on previous study, the incidence rate of PCI-related myocardial injury is 28.7% in UAP patients undergoing PCI. And in our study the expected incidence rate of PCI-related myocardial injury is up to 14.3% in UAP patients undergoing PCI after treatment with low temperature contrast. Moreover, the investigators estimated 10% loss follow-up of these patients in each arm. As a result, a total of 440 UAP patients were required, and with 220 patients per group as a ratio of 1:1 randomization.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesions
* Those who meet the diagnostic criteria of unstable angina pectoris
* New generation drug eluting stent implantation
* Only single coronary artery treated at this time

Exclusion Criteria:

* Those who meet the diagnostic criteria of acute myocardial infarction
* Those who meet the diagnostic criteria of stable angina pectoris
* Patients with cardio-genic shock
* Patients with multiple organ failure
* Patients allergic to contrast
* Patients who can not tolerate dual antiplatelet therapy
* Patients who can't tolerate anticoagulation
* Recently infected patients
* Patients with hepatorenal dysfunction
* Thrombotic lesion of coronary artery
* Chronic total coronary occlusion lesion
* Patients with complex coronary bifurcation requiring two stent strategy
* Severe coronary calcified lesion
* Patients with percutaneous coronary angioplasty
* Patients with directional coronary atherectomy or rotational atherectomy
* Patients with drug coated balloon treatment
* Patients with bioabsorbable vascular scaffold implantation
* Previous percutaneous coronary intervention or coronary artery bypass graft
* Patients with active stage of autoimmune disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence rate of PCI-related myocardial injury in UAP patients 3 days after PCI | 3 days after PCI
  the incidence rate of PCI-related myocardial injury indicated by the changes of myocardial injury biomarkers (such as TNI and CK-MB) in UAP patients between low temperature contrast and room temperature contrast groups

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ye, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (7):
- China (7):
  - The First People's Hospital of Chuzhou, Chuzhou, Anhui
  - MingGuang People's Hospital, Chuzhou, Anhui
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The People's hospital of Yixing, Yixing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moschovitis A, Cook S, Meier B. Percutaneous coronary interventions in Europe in 2006. EuroIntervention. 2010 Jun;6(2):189-94. doi: 10.4244/EIJV7I6A31. PMID 20562067
- [Background] Testa L, Van Gaal WJ, Biondi Zoccai GG, Agostoni P, Latini RA, Bedogni F, Porto I, Banning AP. Myocardial infarction after percutaneous coronary intervention: a meta-analysis of troponin elevation applying the new universal definition. QJM. 2009 Jun;102(6):369-78. doi: 10.1093/qjmed/hcp005. Epub 2009 Mar 13. PMID 19286891